CLINICAL TRIAL: NCT00194961
Title: A Multicenter Study of the Effect of Recombinant Human Growth Hormone on Leptin and Cytokines in Relation to Body Composition in Pediatric Patients With Growth Failure Due to Chronic Kidney Disease (CKD)
Brief Title: Effect of Growth Hormone on Leptin, Cytokines and Body Composition of Children With Growth Failure Due to Chronic Kidney Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding was not approved
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2758s; M2758s
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Growth Failure; Cytokines; leptin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Failure to Thrive | interventions — Growth Hormone

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone

SUMMARY:
Circulating concentrations of cytokines, such as leptin, tumor necrosis factor-alpha and interleukins 1 and 6 are increased in patients with chronic kidney disease (CKD). In light of the increasing recognition that growth hormone receptor signaling involves cytokine pathway activation, the investigators hypothesize that maladaptation of cytokine regulation in chronic kidney disease may underlie growth failure. Secondly, they hypothesize that administration of recombinant human growth hormone (rhGH) will result in growth rate stimulation in pre-pubertal children with growth impairment due to chronic kidney disease by down regulation of the cytokine pathways.

This is a non-randomized open-label study to evaluate the effect of recombinant human growth hormone on biochemical/metabolic and immunologic parameters in relation to body composition pre- and post-recombinant human growth hormone therapy of pre-pubertal growth hormone naive children. The efficacy of recombinant human growth hormone to improve growth velocity in pre-pubertal children with growth failure is a secondary objective. Fifteen children are to be studied over a six month period. Each patient will serve as his/her own control. Six months of growth data prior to study is required.

DETAILED DESCRIPTION:
Hypothesis: The energy cost of growth is increased in experimental CKD. Caloric intake has been shown to correlate with height velocity in children with CKD, and calorie supplementation has been clearly shown to improve height velocity in children on dialysis. However, when energy intake exceeds 75% of the recommended allowance, further growth improvement does not occur. Circulating concentrations of cytokines, such as leptin, tumor necrosis factor-alpha and interleukins 1 and 6 are increased in patients with CKD. In light of the increasing recognition that growth hormone receptor signaling involves cytokine pathway activation, we hypothesize that maladaptation of cytokine regulation in CKD may underlie growth failure. Secondly, we hypothesize that administration of recombinant human growth hormone (rhGH) will result in growth rate stimulation in pre-pubertal children with growth impairment due to CKD by down regulation of the cytokine pathways.

Specific Aims: This investigation's primary objective will be to evaluate biochemical/metabolic, and immunologic parameters in relation to body composition pre- and post-rhGH therapy. The secondary objective is to examine the efficacy of rhGH to improve growth velocity in prepubertal, rhGH naïve, children with growth failure secondary to CKD. The safety of rhGH will be assessed by measuring the above parameters, in addition to identifying if there is an increase in the incidence of slipped capital femoral epiphyses, and an increase in progression of the underlying renal disease.

Methods of Procedure: This is an open-label study to evaluate the efficacy and safety of recombinant human growth hormone in children with chronic kidney disease and growth failure.

The study involves obtaining the following:

1. Medical History and Physical Examination: Subjects will have a complete medical history for any potential conditions/medications, which might affect linear growth, growth velocity, or responsiveness to rhGH. A complete physical examination will be performed, including Tanner Staging, accurate measurement of standing height (or recumbent length, if < 3 years of age) using a stadiometer (in triplicate), weight (in triplicate), blood pressure and funduscopic examination at each referring Center. Anthropometric measurements will be made at the Body Composition Unit at St. Luke's-Roosevelt Medical Center, New York, NY.
2. Routine labs will include a CBC (Hgb/ Hct), BUN, creatinine, liver function studies, and albumin.
3. Bone Age
4. Leptin
5. Cytokines that will be measured include IL-6, TNF alpha, TNFsR, Rp55 (type1), IL-1beta, and IL-1Ra. The ratio of IL-1 to IL-1Ra will be measured as intracellular and extracellular IL-1b compared to extracellular IL-Ra measured in circulation and as produced in vitro, both spontaneously and in response to activation. TNF alpha levels and production both intracellularly and extracellularly will be compared to TNFsRp55 (type 1)
6. Insulin
7. GH-IGF Axis Proteins
8. Body Composition by DXA

During the two years of the study, we anticipate that 15 eligible subjects will receive rhGH at 0.05 mg/kg daily by subcutaneous injection. This estimate of patient enrollment is based upon our preliminary data and our experience with the incidence, age of onset of CKD, and the anticipated change in therapy as some of these patients receive transplants. The dose will be calculated based on the initial weight and will be adjusted as needed every three months according to weight. A parent or legal guardian will administer all doses at home after appropriate training. Following treatment for 6 months and termination from the study, patients who remain eligible due to persistent growth retardation, will receive daily rhGH as standard of care therapy at their institution and their growth rates will be followed. During the course of the study all study subjects will continue medical management and follow-up of their CKD as prescribed by their Pediatric Nephrologist. Subjects may require concomitant medications such as erythropoietin, calcium supplements, sodium bicarbonate/sodium citrate, phosphate binders, calcitriol, and/or antihypertensives as part on their on-going management.

After baseline assessment (Time 0), all study subjects will enter a six-month observation phase. Medical history, physical examination, biochemical studies, creatinine clearance for glomerular filtration rate (GFR), Hgb/Hct, Glucose Tolerance testing (GTT) with insulin measurements, GH-IGF axis proteins, cytokine and leptin studies will be obtained at Time 0, +3 months, and +6 months. At Time 0 and at the end of six months of observation, study subjects will also undergo body composition evaluation (DXA) for a total of two sets of studies. Bone age will be assessed at these time points as well. Each patient will serve as his/her own control at Time 0 for all these measurements. Historical growth data will be obtained back as far as six months, and further, if possible.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal insufficiency as defined by the North American Pediatric Renal Transplant Cooperative Study (NAPRTCS; estimated creatinine clearance < 75 ml/min/1.73 m2 by the Schwartz formula
* Tanner Stage I or II
* Availability of growth data for the preceding 6 months, and growth failure defined as height < 5th percentile for chronological age, and/or SDS score for height more negative than -1.88, and/or height velocity SDS < 0 for six months

Exclusion Criteria:

* Unable or unwilling to adhere to the protocol
* Additional diagnoses that could impair responsiveness to GH, e.g. dwarfism syndromes or significant extra-renal organ disease, e.g. chronic liver disease, diabetes mellitus, AIDS
* Taking medications that influence growth
* Slipped capital femoral epiphysis or avascular necrosis of femoral head
* Constitutional short stature
* Lack of growth potential, e.g. closed epiphysis
* Steroid therapy within previous 3 months
* Known allergy or sensitivity to rhGH
* Previous exposure to a growth hormone product (the patients must be naïve to growth hormone)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Study Completion 2007-12

PRIMARY OUTCOMES:
The primary objective will be to evaluate biochemical/metabolic, and immunologic parameters in relation to body composition. | pre- and post-rhGH therapy

SECONDARY OUTCOMES:
The secondary objective is to examine the efficacy of rhGH to improve growth velocity in prepubertal, rhGH naïve, children with growth failure secondary to CKD.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie L Johnson, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States